CLINICAL TRIAL: NCT00899860
Title: Renal Cell Cancer Tumor Markers
Brief Title: Gene Expression in Normal Tissue and Tumor Tissue From Patients Who Have Undergone Surgery For Kidney Cancer
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000550079; P30CA012197 (NIH); CCCWFU-89A03; CCCWFU-GB03-404
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2012-06

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with renal cell cancer

SUMMARY:
RATIONALE: Studying the genes and proteins expressed in tissue samples from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This laboratory study is evaluating gene and protein expression in normal tissue and tumor tissue from patients who have undergone surgery for kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the expression levels of novel genes and proteins (HFARP, HAMGR28, HE9NG77) in frozen normal tissue and tumor tissue samples from patients who have undergone nephrectomy for renal cell cancer.
* Correlate gene and protein expression levels with disease stage, tumor size, and pathology reports (e.g., cell type, grade, and tissue architecture) in order to evaluate the rate of gene and protein expression as targets for future therapeutic interventions.

Secondary

* Compare proteomic screening of potential biomarkers using existing plasma and/or urine samples from patients with renal cell cancer or breast cancer stored in the CCCWFU Tumor Tissue Core with tissue samples from patients enrolled in this study.

OUTLINE: Normal and tumor tissue collected from patients who have undergone nephrectomy and diagnostic and therapeutic intervention for renal cell cancer is analyzed for histopathological expression and compared to normal kidney cells by northern blot. Tissue samples are evaluated by RNA and protein extraction and analyzed by gel electrophoresis, blotting, and phosphor-imaging for induction or suppression of genes and protein levels. These data are correlated with clinical stage, tumor size, and histopathological grade and architecture of the patient's disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell cancer
* Clinical staging (if available)
* Underwent nephrectomy for renal cell cancer

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those wiht histologically confirmed renal cell cancer who have underwent nephrectomy for renal cell cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2003-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Expression levels of novel genes and proteins (HFARP, HAMGR28, HE9NG77) in frozen normal tissue and tumor tissue | day 1
Correlation of gene and protein expression levels with disease stage, tumor size, and pathology reports | day 1

SECONDARY OUTCOMES:
Comparison of proteomic screening of potential biomarkers using plasma and/or urine samples from patients with renal cell cancer or breast cancer stored in the CCCWFU Tumor Tissue Core with tissue samples from patients enrolled in this study | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Torti, MD, MPH, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States